CLINICAL TRIAL: NCT00574041
Title: An Open-Label Study to Examine the Difference in Tolerability Associated With Titration Of Dose on Initiation of Avonex therapY (TODAY)
Brief Title: How Side Effects of Avonex Are Affected by Gradually Increasing to Full Dose vs Starting at Full Dose
Acronym: TODAY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to poor recruitment
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUS-8002
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Avonex; side effects; flu like symptoms
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): titrated dose of Avonex
  Interventions: Drug: Interferon beta-1a
- 2 (Active Comparator): full dose Avonex
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Interferon beta-1a — injected, once a week
  Other Names: Avonex

SUMMARY:
This study is to find out if starting at low dose Avonex and slowly increasing to full dose will improve flu like symptoms as a side effect of Avonex treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically-definite relapsing-remitting multiple sclerosis

Exclusion Criteria:

* Any Product Information-specified contraindications to interferon-beta therapy, or other medical factors which, in the opinion of the investigator, make the subject unsuitable for interferon-beta therapy
* Use of AVONEX, but not other interferon therapies, in the 3 months prior to randomisation into the study
* A clinically significant infectious illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days prior to randomisation.
* History of seizure in the 3 months prior to randomisation
* History of suicidal ideation or severe depression within the 3 months prior to randomisation.
* Other inclusion and exclusion criteria may apply per study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To assess the mean severity of episodes of FLS during the 4 week titration phase | 4 weeks

SECONDARY OUTCOMES:
To assess the mean severity and duration of FLS episodes in post-titration phase | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — Biogen
Locations (1):
- Coordinating Research Site, Malvern, Victoria, Australia